CLINICAL TRIAL: NCT02436018
Title: Safety and Efficacy Evaluation of The Nasopharyngeal Airway Embedded With Jet Ventilation Catheter(WEI NASAL JET) Applied for The Sedation of Outpatient Upper Gastrointestinal Endoscopy
Brief Title: WEI NASAL JET for The Sedation of Outpatient Upper Gastrointestinal Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pudong New Area People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, diansan su, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RenJiH-20150308
Record Dates: First submitted 2015-04-26; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Peptic Ulcer; Gastric Cancer; Esophagus Cancer; Oesophagitis; Hypoxia
Keywords: Sedation; Low pulse oximetry; Upper gastrointestinal endoscopy; WEI NASAL JET
MeSH Terms: conditions — Peptic Ulcer; Stomach Neoplasms; Esophageal Neoplasms; Esophagitis; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): Oxygen(2L/min) supplied with nasal catheter
- Nasopharyngeal airway group (Experimental): Oxygen(2L/min) supplied directly through WEI NASAL JET without jet ventilator
  Interventions: Device: Nasopharyngeal airway without jet ventilator
- WEI NASAL JET group (Experimental): Oxygen supplied through WEI NASAL JET with a manual jet ventilator
  Interventions: Device: WEI NASAL JET

INTERVENTIONS:
Device: WEI NASAL JET — Oxygen is supplied through WEI NASAL JET by a manual jet ventilator
  Other Names: Nasopharyngeal airway embedded with jet ventilation catheter
  Arms: WEI NASAL JET group
Device: Nasopharyngeal airway without jet ventilator — Oxygen is supplied directly through WEI NASAL JET without jet ventilator
  Arms: Nasopharyngeal airway group

SUMMARY:
Low pulse oximetry is the most common adverse events during sedation for upper gastrointestinal endoscopy. The main reason is the glossoptosis after sedation. In present study a new designed nasopharyngeal airway embedded with jet ventilation catheter(WEI NASAL JET) will be utilized in order to reduce the hypoxia. At the same time the safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing upper gastrointestinal endoscopy
* age over 18 years old
* Signed informed consent form

Exclusion Criteria:

* a blood coagulation dysfunction or have a tendency of nose bleeding
* a clear diagnosis of heart disease (heart failure, angina, myocardial infarction, arrhythmia, etc.)
* a clear diagnosis of lung disease (asthma, chronic obstructive pulmonary disease, pulmonary embolism, pulmonary edema, lung cancer)
* pregnant
* liver disease
* kidney disease
* increase in intracranial pressure
* emergency operation
* multiple trauma
* American Society of Anesthesiologists (ASA) Physical Status classification above IV
* with mouth, nose and throat infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Low pulse oximetry incidence | Patients will be followed for the duration of hospital stay, an expected average of 2 hours

SECONDARY OUTCOMES:
Other adverse events | Patients will be followed for the duration of hospital stay, an expected average of 2 hours
  The adverse events according to the Adverse event reporting tool of the world SIVA International Sedation Task Force during upper gastrointestinal endoscopy will be recorded. Adverse events associated with jet ventilation also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (3):
- China (3):
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Renji hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Qin Y, Li LZ, Zhang XQ, Wei Y, Wang YL, Wei HF, Wang XR, Yu WF, Su DS. Supraglottic jet oxygenation and ventilation enhances oxygenation during upper gastrointestinal endoscopy in patients sedated with propofol: a randomized multicentre clinical trial. Br J Anaesth. 2017 Jul 1;119(1):158-166. doi: 10.1093/bja/aex091. PMID 28974061